CLINICAL TRIAL: NCT02075437
Title: Feelings and Body Investigators (FBI): Interoceptive Exposure for Child Abdominal Pain
Brief Title: Feeling and Body Investigators for Pediatric Abdominal Pain
Acronym: FBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00043556; MH097959 (Other Grant/Funding Number: Federal Identifier)
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Results first posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Functional Abdominal Pain
Keywords: Functional Abdominal Pain, Children; Finding a treatment or intervention for children

ARMS (1):
- Functional Abdominal Pain (FAP) (Experimental): To access (FAP) subjects will participate in: 10 therapy sessions; and the following treatments: 1) identify strategies with unique patterns of neural circuit maturation associated with early visceral pain on the gut-brain axis: 2) adapt acceptance-based behavioral strategies used to address psychopathology in older children to younger children; and 3) incorporate caregivers as role models and facilitators based on attachment research.
  Interventions: Behavioral: Feeling and Body Investigators with Functional Abdominal Pain; Behavioral: Treatment Strategies

INTERVENTIONS:
Behavioral: Feeling and Body Investigators with Functional Abdominal Pain — Investigator's ten session intervention trains children to be "Feeling and Body Investigators". Half of the sessions will be done in clinic and half at home via web-camera to facilitate generalization. During the treatment child/caregiver dyads will 1) gather body clues (Learn), 2) investigate (Experience: perform interoceptive mystery missions to explore a body sensation), 3) organize body clues (Contextualize: recall other context that evoke similar sensations), and 4) go on increasingly daring missions (Challenge: decrease avoidance and safety behaviors).
  If successful, young children with FAP who complete the FBI early intervention will learn to experience changes in the viscera as fun and fascinating, rather than scary, and will develop new capacities for pain management, adaptive functioning, and emotion regulation.
  Other Names: Ten Session Therapy for Young Children with Functional Abdominal Pain
Behavioral: Treatment Strategies — 1. identify strategies with unique patterns of neural circuit maturation associated with early visceral pain on the gut-brain axis:
  2. adapt acceptance-based behavioral strategies used to address psychopathology in older children to younger children;
  3. incorporate caregivers as role models and facilitators based on attachment research.

SUMMARY:
This study will provide tools to develop and pilot an intervention for Functional Abdominal Pain (FAP) using a ten session intervention with children ages 5-8. Investigators will train the subjects to be "Feeling and Body Investigators". During treatment phases the following will occur 1) gather clues (learn), 2) investigate (experience: perform interoceptive mystery missions to explore a body sensation), 3) organize body clues (contextualize: recall other contexts that evoke similar sensations), and 4) go on increasingly daring missions (challenge: decrease avoidance and safety behaviors). The FBI intervention will be developed and refined in 28 child-caregiver dyads during the current R21 phase. In the R33 phase investigators will randomize 100 subjects with FAP to FBI or an active control group in order to conduct a pilot-test of the feasibility, acceptance, and clinical significance of FBI. Young children with FAP who complete the FBI early intervention will learn to experience changes in the viscera as fun and fascinating, rather than scary, and will develop new capacities for pain management, adaptive functioning, and emotion regulation. For the R21 Phase (assessing initial feasibility) investigators hypothesize that ≥ 80% of participants enrolled in FBI will complete treatment and that ≥ 80% of participants will complete home-based practice assignments.

ELIGIBILITY:
Inclusion Criteria:

* Child is between 60 and 107 months old.
* Parent/legal guardian is present at the clinic visit who speaks English
* Child screens positive for recurrent abdominal pain by having: 1) 8 episodes of abdominal pain over 2 months (based on Rome III criteria), or 2) 2 or more episodes of abdominal pain which are causing an incapacity greater than or equal to 25% of the time in the past two months).
* Based on pediatric medical assessment, child meets criteria for functional abdominal pain (FAP) based on absence of other organic causes of recurrent abdominal pain.
* Consent given by caregiver and assent by child to participate.
* Presence of internet access, including that accessed by cell phone with video capabilities.

Exclusion Criteria:

* The index child being known to have mental retardation (IQ < 70) or other pervasive developmental disorders.
* Subject has a sibling who is already enrolled in our study. ***Possible Exclusion***
* Parent/ guardian who would be participating in the study is pregnant.

Ages: 60 Months to 107 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Zucker, PhD, Principal Investigator — Director, Duke Center for Eating Disorders, Professor; Helen Egger, MD, Principal Investigator — Head, Division of Child and Adolescent Psychiatry, Associate Professor
Locations (2):
- United States (2):
  - Duke University Young Child Lab at Brightleaf Square, Durham, North Carolina
  - Duke Children's Primary Care Picket Road, Durham, North Carolina

REFERENCES:
- [Derived] Zucker N, Mauro C, Craske M, Wagner HR, Datta N, Hopkins H, Caldwell K, Kiridly A, Marsan S, Maslow G, Mayer E, Egger H. Acceptance-based interoceptive exposure for young children with functional abdominal pain. Behav Res Ther. 2017 Oct;97:200-212. doi: 10.1016/j.brat.2017.07.009. Epub 2017 Jul 29. PMID 28826066

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Caregiver-child dyads were enrolled to examine the acceptability and feasibility of a new treatment for child abdominal pain. Caregiver-child dyads were enrolled in the study protocol and both involved in treatment sessions.
Groups:
- Feeling and Body Investigators (FBI) Caregiver-Child Dyads: Feeling and Body Investigators (FBI) is a 10-session intervention to treat children with functional abdominal pain. The treatment contains the following components: 1) We aim to reduce fearful perceptions of somatic and visceral sensations by linking sensations to playful characters. In sessions organized by theme (e.g., the Eats), children build curious reactions to things they notice in their bodies using funny cartoon characters used to teach them the meaning of different sensations (e.g. Betty Butterfly for gut butterflies of anxiety). 2) Children perform interoceptive exposure activities designed to demonstrate how smart and tough the body is in responding to different demands (e.g., seeing how fast a child can run even if they feel uncomfortable). 3) Children learn to link body sensations to meanings and actions. Using a Body Clues Worksheet, children figure out what they were feeling, what their feeling was telling them, and try out different ways to respond to the messages of their body to see what happens. 4) Families design investigations to help them face challenging situations (e.g. devising a plan to run around at recess to try to get all their gas out and see what happens to their abdominal pain after recess). If successful, kids with FAP who complete treatment will learn to experience body sensations as fun and fascinating, rather than scary, and develop new capacities for pain management, increase adaptive functioning, and enhance interoceptive responsivity.
Period: Overall Study
Arm/Group | Feeling and Body Investigators (FBI) Caregiver-Child Dyads
Started | 28 (In our participant data flow during this phase of the clinical trial there were a total of 28 caregiver-child dyads the started that study)
Completed | 22 (In our participant data flow during this phase of the clinical trial there were a total of 22 caregiver-child dyad that completed treatment sessions)
Not Completed | 6
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics were not collected from caregivers.
Groups:
- Feeling and Body Investigators (FBI) Caregiver-Child Dyads - Children: Feeling and Body Investigators (FBI) is a 10-session intervention to treat children with functional abdominal pain. The treatment contains the following components: 1) We aim to reduce fearful perceptions of somatic and visceral sensations by linking sensations to playful characters. In sessions organized by theme (e.g., the Eats), children build curious reactions to things they notice in their bodies using funny cartoon characters used to teach them the meaning of different sensations (e.g. Betty Butterfly for gut butterflies of anxiety). 2) Children perform interoceptive exposure activities designed to demonstrate how smart and tough the body is in responding to different demands (e.g., seeing how fast a child can run even if they feel uncomfortable). 3) Children learn to link body sensations to meanings and actions. Using a Body Clues Worksheet, children figure out what they were feeling, what their feeling was telling them, and try out different ways to respond to the messages of their body to see what happens. 4) Families design investigations to help them face challenging situations (e.g. devising a plan to run around at recess to try to get all their gas out and see what happens to their abdominal pain after recess). If successful, kids with FAP who complete treatment will learn to experience body sensations as fun and fascinating, rather than scary, and develop new capacities for pain management, increase adaptive functioning, and enhance interoceptive responsivity.
Arm/Group | Feeling and Body Investigators (FBI) Caregiver-Child Dyads - Children
Number analyzed (Participants) | 28
Age, Continuous [Mean (Full Range); unit: years] | 7.04 [5.02 to 9.30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 21
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Complete Treatment
Description: Treatment in this study refers to 10 treatment sessions (2 over cell phone video chat from the subject's home and 8 in the investigator's lab) using an acceptance-based behavioral treatment for children 5 through 9 years old with impairing functional abdominal pain. This intervention is rooted in a biopsychosocial framework incorporating advances in neurodevelopment, behavioral learning theory, and attachment theory.
Time Frame: 1.5 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Feeling and Body Investigators (FBI) Caregiver-Child Dyads
Number analyzed (Participants) | 28
Participants | 22

2. Primary Outcome: Number of Participants Completing Homework Assignment
Description: Enrollees will engage in assigned home-based practice sessions for at least nine of the ten treatment weeks. Completion of assigned practice sessions within a given week is defined as success.
Time Frame: 1.5 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Feeling and Body Investigators (FBI) Caregiver-Child Dyads
Number analyzed (Participants) | 28
Participants | 15

ADVERSE EVENTS:
Time Frame: 1.5 years
Description: Only children were monitored for adverse events. Caregivers and children provided any info related to adverse events throughout the duration of their involvement in this clinical trial.
Arm/Group | Feeling and Body Investigators (FBI) Caregiver-Child Dyads - Children
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/37/NCT02075437/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/37/NCT02075437/SAP_001.pdf
  • Informed Consent Form (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/37/NCT02075437/ICF_002.pdf